CLINICAL TRIAL: NCT01118169
Title: Examining the Relationship Between Personal Values, Interpersonal Needs, and Suicidal Ideation in a Veteran Population
Brief Title: Personal Values, Interpersonal Needs, and Suicidal Ideation in a Veteran Population
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nazanin H. Bahraini, Research/Clinical Psychologist, VA Eastern Colorado Health Care System
Other Study IDs: COMIRB 09-0523
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Suicide Prevention
Keywords: Personal values; Suicidal thoughts
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veterans

SUMMARY:
The primary aim of this study is to examine the relationship between personal values and suicidal thoughts in a sample of U.S. Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving care through the Denver VA Medical Center Behavioral Health Interdisciplinary Team
* Over the age of 18
* Willing to travel to the Denver VAMC to complete assessment measures.
* Provide informed consent to participate

Exclusion Criteria:

* Inability to adequately respond to questions regarding the informed consent procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans receiving behavioral health services within the Denver VA Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Beck Scale for Suicide Ideation | One time
  Questionnaire that assesses suicidal thoughts

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, Ph.D., Study Director — VA Eastern Colorado Health Care System
Locations (1):
- Denver VA Medical Center, Denver, Colorado, United States